CLINICAL TRIAL: NCT06677346
Title: Investigating the Relationship Between Parity and Respiratory Muscle Strength in Women.
Brief Title: Parity and Respiratory Muscle Strength in Women
Status: Recruiting | Type: Observational
Sponsor: Medipol University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); Istanbul Kültür University (Other)
Responsible Party: Principal Investigator, Imge NAS, Lecturer, Istanbul Kültür University
Other Study IDs: İK-2023-02
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Respiratory Muscle Strength; Parity; Core Stability; Woman

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Nulliparous: Women who have never given birth
- Primiparous: Women who have given birth once
- Multiparous: Women who have given birth multiple times

SUMMARY:
The aim of this study is to investigate the relationship between parity and respiratory muscle strength in women.

DETAILED DESCRIPTION:
In normal anatomical structure, there is myofascial continuity between the diaphragm, abdominal muscles and pelvic floor muscles. In addition to this anatomical unity, when the diaphragm muscle descends with inhalation, the pelvic floor muscle moves caudally, allowing breathing to encounter less resistance; the opposite occurs during exhalation.

Pregnancy and childbirth create anatomical and physiological changes in the female body. As a result of the growing uterus, the diaphragm moves upwards, while the pelvic floor muscles become depressed as intra-abdominal weight increases. On the other hand, it is thought that increased ligament laxity is responsible for changes in the body's muscle structure, especially in the lower body. Considering these pregnancy-related changes, the functions of these interrelated muscle groups may be affected and synergistic movements in the woman's body may be disrupted after pregnancy.

The aim of this study is to examine whether the anatomical structures affected during pregnancy have permanent effects on respiratory muscle strength and core muscles after birth. Volunteers who agree to participate in the study will be divided into groups according to their birth counts and respiratory and core muscles will be evaluated using objective methods.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-45 years old
* Being female

Exclusion Criteria:

* Having a body mass index of ≥30 kg/m2
* History of cardiovascular, neurological, pulmonary disease
* Being receiving active cancer treatment
* Having a history of lumbar surgery
* History of smoking
* Being a licensed athlete

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The participant group of the research will consist of women between the ages of 20-45 and participation will be based on volunteering.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Respiratory Muscle Strength/ maximal inspiratory pressure (MIP) | On the day of enrollment
  Participants' maximal inspiratory pressure (MIP) measurements will be evaluated using the COSMED Pony FX spirometry device according to American Thoracic Society/European Respiratory Society standards.
Respiratory Muscle Strength/maximal expiratory pressure (MEP) | On the day of enrollment
  Participants' maximal expiratory pressure (MEP) measurements will be evaluated using the COSMED Pony FX spirometry device according to American Thoracic Society/European Respiratory Society standards.

SECONDARY OUTCOMES:
Pressure Biofeedback Unite | On the day of enrollment
  Core muscle stabilization will be measured with The Stabilizer Pressure Biofeedback Unit. Individuals are asked to lie down in the supine and prone positions. After the pressure cell of the instrument is placed with reference to the Anterior superior iliac spines (ASIS) and Posterior superior iliac spines (PSIS), the subjects are asked to perform a drawing-in maneuver. The contraction that can be sustained for 10 seconds is recorded in mmHg.
Trunk Muscle Endurance Tests | On the day of enrollment
  The endurance of the trunk flexor, trunk extensor and lateral flexor muscles is evaluated by recording the maximum time that the person can maintain the test position.
Physical Activity Level | On the day of enrollment
  Individuals' physical activity levels will be questioned with the International Physical Activity Questionnaire (IPAQ) Short Form. It is a 7-item scale. Physical activity levels are classified into 3 categories according to the scores obtained by multiplying the duration, frequency and MET values of the physical activities that the participants participated in within 7 days and for at least 10 minutes. Accordingly, <600 MET - min/week is defined as inactive, 600 - 3000 MET - min/week low, and >3000 MET - min/week is defined as sufficient physical activity level.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Kultur University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No